CLINICAL TRIAL: NCT07011316
Title: Subclinical Assessment and Monitoring of Lymphatic System Function in Oncology Patients as Part of Physiotherapeutic Prevention of Limb Lymphoedema
Brief Title: Subclinical Monitoring of Lymphatic Function in Oncology Patients for Lymphoedema Prevention (ONCOLYMPH)
Acronym: ONCOLYMPH
Status: Recruiting | Type: Observational
Sponsor: The Greater Poland Cancer Centre (Other)
Collaborators: Poznan University of Physical Education (Other)
Responsible Party: Sponsor
Other Study IDs: ONCOLYMPH
Record Dates: First submitted 2025-04-28; First posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: Lymphoedema
Keywords: Lymphoedema; Cancer; Prevention; bioimpedance spectroscopy
MeSH Terms: conditions — Lymphedema; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Main patient cohort: * 150 women with malignant tumours of the urinary and genital systems
  * 150 men with malignant tumours of the urinary and genital systems
  * 150 patients with malignant tumours of the nipple (breast)
  * 150 patients with malignant tumours of the nipple (breast) and malignant tumours of the urinary and genital systems treated with brachytherapy

SUMMARY:
Lymphoedema, a chronic condition caused by the accumulation of protein-rich fluid in the intercellular spaces due to impaired lymphatic function, is a common complication in cancer patients. It can lead to visible swelling, discomfort, and mobility issues, but most frequently affects the limbs. This condition not only impacts patients physically but also has significant psychological consequences, including reduced quality of life, social stigma, and challenges with returning to daily activities.

Oncology patients are particularly at risk for developing lymphoedema due to factors such as lymphadenectomy, radiotherapy, and extensive surgical procedures. Up to 30% of breast cancer survivors develop lymphoedema, and it is also a common complication in patients treated for other cancers, such as those involving the cervix, vulva, prostate, and bladder. Despite the importance of early detection, diagnostic tools for assessing lymphatic dysfunction are often specialised and not suitable for routine screening in clinical practice.

The primary goal of this study is to explore the early signs of lymphatic dysfunction in cancer patients before evident clinical symptoms, with the aim of identifying individuals at risk of developing lymphoedema. This will provide valuable information that could guide early interventions and preventive measures to reduce the severity or even prevent the onset of lymphoedema. By focusing on early, subclinical dysfunction, the study seeks to contribute to improving both the clinical management of lymphatic complications and the overall quality of life for oncology patients. Regular monitoring and timely physiotherapy interventions could play a key role in enhancing recovery outcomes and reducing the long-term impact of lymphoedema.

DETAILED DESCRIPTION:
Lymphoedema is a chronic condition characterised by an increase in body volume due to the accumulation of protein-rich fluid and cellular debris in the interstitial spaces, resulting from impaired lymphatic vessel function. It can affect various areas of the body, such as the external genitalia, abdomen, and face, but most commonly occurs in the limbs, leading to visible swelling and associated discomfort.

The main risk factors for lymphoedema include lymphadenectomy, radiotherapy, extensive surgical procedures, and obesity. Oncology patients frequently experience this condition as a complication of cancer treatment. According to data from the World Health Organization, up to 30% of breast cancer survivors develop lymphoedema. It is also a common complication in patients treated for other cancers usually as a result of surgical removal of lymph nodes or radiotherapy that damages structures of the lymphatic system (cancer of the: cervix ~ 30%; vulva ~ 27%; sarcoma ~ 27%; penis ~ 25% melanoma ~ 23%; prostate ~ 18%; bladder ~ 15%; testes: ~ 10%).

Lymphoedema diagnosis is based on clinical examination and the exclusion of other causes, primarily chronic venous insufficiency and thrombosis. Standard diagnostic methods like lymphoscintigraphy and indocyanine green (ICG) dye lymphography require specialised equipment and conditions, making them less suitable for routine screening to assess lymphatic damage and the risk of lymphoedema development.

Individuals affected by lymphoedema experience not only physical symptoms such as inflammation and mobility issues but also psychological effects, including reduced quality of life, social stigma, and challenges in returning to work. According to the International Society of Lymphology (ISL), lymphoedema treatment should be interdisciplinary, incorporating a comprehensive range of therapeutic approaches such as pharmacotherapy, surgery, multi-layer compression, pneumatic compression, manual lymphatic drainage, and specialised exercises to enhance lymph flow. As the course of treatment is prolonged and the results are not fully satisfactory, methods and programmes to prevent the formation and development of lymphoedema are of particular importance, both clinically and economically.

Regular monitoring of lymphatic system function in oncology patients and the early implementation of physiotherapy can significantly reduce the risk of lymphoedema or limit its severity, ultimately improving patients' quality of life and recovery outcomes.

Purpose of the research: The aim of the project is to assess early - subclinical peripheral lymphatic system dysfunction resulting from various treatment modalities (surgery, radiotherapy, brachytherapy) in oncology patients. The study will include patients with breast cancer, malignant urinary and genital cancers, both treated surgically and/or with brachytherapy. Recruited patients' body composition will be assessed using non-invasive technology of spectroscopic bioimpedance analysis (BIA) with a body composition analyser - SOZO® Digital Health Platform apparatus. Measurements will be taken three times: (1) before the start of treatment on admission to the hospital, (2) after the applied treatment before the patient is discharged, and (3) at the standard follow-up visit two/three months after the end of treatment in the hospital. The assessment of the efficiency of the lymphatic system provides information on the appropriateness of taking preventive measures to prevent the development of lymphoedema of the limbs.

ELIGIBILITY:
Inclusion Criteria:

* admission to the Greater Poland Cancer Centre for treatment in one of the departments participating in the study,
* age ≥ 18 years,
* ability to balance independently in a standing position for 30 seconds,
* obtaining the patient's written informed consent to participate in the study.

Exclusion Criteria:

* age ≤ 18 years,
* cardiac arrhythmia,
* pacemakers or other implanted electronic devices,
* history of external defibrillation,
* pregnancy,
* critical limb ischaemia,
* advanced heart failure (NYHA III and IV0),
* symptoms of deep vein thrombosis,
* uncompensated heart, kidney or thyroid failure,
* peripheral nerve damage,
* presence of psychiatric disorders that preclude informed consent or limit appropriate co-operation of the patient,
* lack of informed consent from the patient to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals affected by lymphoedema experience not only physical symptoms such as inflammation and mobility issues but also psychological effects, including reduced quality of life, social stigma, and challenges in returning to work.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
L-Dex ratio | Time Frame: Metrics assessed at baseline (within two weeks before treatment), after treatment (up to 2 weeks after completing treatment/intervention), and during follow-up (up to 8 weeks ± 2 weeks after completing treatment/intervention)
  The assessment of lymphoedema will be performed using non-invasive technology of spectroscopic bioimpedance analysis (BIA) with a body composition analyser - SOZO® Digital Health Platform apparatus and measured as L-Dex parameter. L-Dex ratio will be calculated by dividing the bioimpedance reading of the affected limb by the bioimpedance reading of the unaffected limb.

SECONDARY OUTCOMES:
BMI | Time Frame: Metrics assessed at baseline (within two weeks before treatment), after treatment (up to 2 weeks after completing treatment/intervention), and during follow-up (up to 8 weeks ± 2 weeks after completing treatment/intervention)
  Body Mass Index; weight in kilograms (kg) and height in meter (m) will be combined to report BMI in kg/m^2. The parameters will be measured using spectroscopic bioimpedance analysis (BIA) with a body composition analyser - SOZO® Digital Health Platform apparatus.
Percent body fat | Time Frame: Metrics assessed at baseline (within two weeks before treatment), after treatment (up to 2 weeks after completing treatment/intervention), and during follow-up (up to 8 weeks ± 2 weeks after completing treatment/intervention)
  Body fat mass in kilograms (kg) and weight in kilograms (kg) will be combined to report Percent body fat in kg/kg*100 (%). The parameters will be measured using spectroscopic bioimpedance analysis (BIA) with a body composition analyser - SOZO® Digital Health Platform apparatus.
Percent body water | Time Frame: Metrics assessed at baseline (within two weeks before treatment), after treatment (up to 2 weeks after completing treatment/intervention), and during follow-up (up to 8 weeks ± 2 weeks after completing treatment/intervention)
  Total body water mass in kilograms (kg) and weight in kilograms (kg) will be combined to report Percent total body water in kg/kg*100 (%). The parameters will be measured using spectroscopic bioimpedance analysis (BIA) with a body composition analyser - SOZO® Digital Health Platform apparatus.

CONTACTS AND LOCATIONS:
Overall Officials: Janusz Doś, PT, PhD, Principal Investigator — The Greater Poland Cancer Centre
Locations (1):
- The Greater Poland Cancer Centre, Poznan, Greater Poland Voivodeship, Poland

REFERENCES:
- [Background] Kilgore LJ, Korentager SS, Hangge AN, Amin AL, Balanoff CR, Larson KE, Mitchell MP, Chen JG, Burgen E, Khan QJ, O'Dea AP, Nye L, Sharma P, Wagner JL. Reducing Breast Cancer-Related Lymphedema (BCRL) Through Prospective Surveillance Monitoring Using Bioimpedance Spectroscopy (BIS) and Patient Directed Self-Interventions. Ann Surg Oncol. 2018 Oct;25(10):2948-2952. doi: 10.1245/s10434-018-6601-8. Epub 2018 Jul 9. PMID 29987599
- [Background] da Silva Tozzo FCB, Sarri AJ, Pirola WE, da Silva UBC, de Oliveira MA, de Padua Souza C, da Costa Vieira RA. Evaluation of upper limb lymphoedema and diagnostic accuracy of bioimpedance spectroscopy. A comprehensive validation in a Brazilian population. Ecancermedicalscience. 2023 Dec 18;17:1649. doi: 10.3332/ecancer.2023.1649. eCollection 2023. PMID 38419858
- [Background] Shah C, Whitworth P, Valente S, Schwarz GS, Kruse M, Kohli M, Brownson K, Lawson L, Dupree B, Vicini FA. Bioimpedance spectroscopy for breast cancer-related lymphedema assessment: clinical practice guidelines. Breast Cancer Res Treat. 2023 Feb;198(1):1-9. doi: 10.1007/s10549-022-06850-7. Epub 2022 Dec 24. PMID 36566297
- [Background] Whitworth PW, Shah C, Vicini F, Cooper A. Preventing Breast Cancer-Related Lymphedema in High-Risk Patients: The Impact of a Structured Surveillance Protocol Using Bioimpedance Spectroscopy. Front Oncol. 2018 Jun 12;8:197. doi: 10.3389/fonc.2018.00197. eCollection 2018. PMID 29946531
- [Background] Torres Lacomba M, Yuste Sanchez MJ, Zapico Goni A, Prieto Merino D, Mayoral del Moral O, Cerezo Tellez E, Minayo Mogollon E. Effectiveness of early physiotherapy to prevent lymphoedema after surgery for breast cancer: randomised, single blinded, clinical trial. BMJ. 2010 Jan 12;340:b5396. doi: 10.1136/bmj.b5396. PMID 20068255
- [Background] Stuiver MM, ten Tusscher MR, Agasi-Idenburg CS, Lucas C, Aaronson NK, Bossuyt PM. Conservative interventions for preventing clinically detectable upper-limb lymphoedema in patients who are at risk of developing lymphoedema after breast cancer therapy. Cochrane Database Syst Rev. 2015 Feb 13;2015(2):CD009765. doi: 10.1002/14651858.CD009765.pub2. PMID 25677413
- [Background] Rio-Gonzalez A, Molina-Rueda F, Palacios-Cena D, Alguacil-Diego IM. Living with lymphoedema-the perspective of cancer patients: a qualitative study. Support Care Cancer. 2018 Jun;26(6):2005-2013. doi: 10.1007/s00520-018-4048-x. Epub 2018 Jan 12. PMID 29330708
- [Background] Ridner SH, Dietrich MS, Boyages J, Koelmeyer L, Elder E, Hughes TM, French J, Ngui N, Hsu J, Abramson VG, Moore A, Shah C. A Comparison of Bioimpedance Spectroscopy or Tape Measure Triggered Compression Intervention in Chronic Breast Cancer Lymphedema Prevention. Lymphat Res Biol. 2022 Dec;20(6):618-628. doi: 10.1089/lrb.2021.0084. Epub 2022 Jan 28. PMID 35099283
- [Background] Park JH, Lee WH, Chung HS. Incidence and risk factors of breast cancer lymphoedema. J Clin Nurs. 2008 Jun;17(11):1450-9. doi: 10.1111/j.1365-2702.2007.02187.x. PMID 18482142
- [Background] Naczk A, Dos J, Gorska-Dos M, Sibilski R, Gramza P, Gajewska E, Naczk M. Relationship between Viscoelastic Properties of Tissues and Bioimpedance Spectroscopy in Breast-Cancer-Related Lymphedema. J Clin Med. 2022 Feb 26;11(5):1294. doi: 10.3390/jcm11051294. PMID 35268385
- [Background] Box RC, Reul-Hirche HM, Bullock-Saxton JE, Furnival CM. Physiotherapy after breast cancer surgery: results of a randomised controlled study to minimise lymphoedema. Breast Cancer Res Treat. 2002 Sep;75(1):51-64. doi: 10.1023/a:1016591121762. PMID 12500934